CLINICAL TRIAL: NCT04902378
Title: Closed-loop Insulin Delivery by Glucose Responsive Computer Algorithms In Type 1 Diabetes Pregnancies (CIRCUIT)
Brief Title: Closed-loop Insulin Delivery In Type 1 Diabetes Pregnancies (CIRCUIT)
Acronym: CIRCUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Lois Donovan, MD, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-1266
Record Dates: First submitted 2021-04-28; First posted 2021-05-26 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus; Pregnancy Related; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases
Keywords: Type 1 diabetes, pregnancy, closed-loop, clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tandem t:slim X2 insulin pump with Control IQ technology plus CGM (Experimental): Participants randomized to the intervention group will be fitted with the Tandem t:slim X2 insulin pump with Control IQ technology and Dexcom G6 Continuous Glucose Monitor.
  Interventions: Device: Tandem t:slim X2 insulin pump with Control IQ technology
- Standard insulin delivery (multiple daily injections (MDI) or pump) and CGM (No Intervention): Participants randomized to the control group will be fitted with the Dexcom G6 Continuous Glucose Monitor. They will continue to use standard insulin delivery (MDI or pump) and CGM.

INTERVENTIONS:
Device: Tandem t:slim X2 insulin pump with Control IQ technology — The intervention group will be fitted with the Tandem t:slim X2 insulin pump with Control IQ technology during pregnancy.
  Arms: Tandem t:slim X2 insulin pump with Control IQ technology plus CGM

SUMMARY:
This trial will assess the efficacy of the Tandem t:slim X2 insulin pump with Control IQ technology compared with standard insulin delivery plus CGM in pregnant women with type 1 diabetes.

DETAILED DESCRIPTION:
Pregnant women with type 1 diabetes (T1D) require normal or near normal glucose in order to reduce the risks of birth defects, stillbirth, increased birthweight, neonatal hypoglycemia, neonatal death, preterm delivery and preeclampsia. Reducing maternal glucose is extremely difficult due to an increased risk of maternal hypoglycemia. Only 14% of T1D pregnancies achieve pregnancy guideline recommended glucose control, leading to complications related to high maternal glucose exposure in roughly half of newborns.

Maintaining recommended maternal glucose levels during pregnancy reduces the risk of adverse neonatal outcomes to those similar in pregnancies unaffected by T1D. Most insulin pumps in use today are open-loop systems, which means that the user must program the pump to deliver a pre-set amount of insulin. These insulin delivery methods (MDI and open-loop pumps) are usually inadequate to achieve the optimal glucose control necessary for T1D pregnancies and they impart a large time, effort and emotional burden.

Closed-loop systems have been found to be effective in improving glucose control outside of pregnancy when studied in children and adults. A new hybrid closed-loop system, the Tandem t:slim X2 insulin pump with Control IQ technology, recently became commercially available. Trials have demonstrated the efficacy of the Control IQ algorithm for non-pregnant adults and children. Pregnant women were not included in these trials.

The investigators propose the first randomized controlled trial to evaluate the Tandem t:slim X2 insulin pump with Control IQ technology versus standard insulin delivery (MDI or pump) and CGM in pregnant women with T1D. In this trial, the investigators will assess the efficacy of the Tandem t:slim X2 insulin pump with Control IQ technology compared with standard insulin delivery plus CGM in pregnant women with type 1 diabetes.

We are grateful to Tandem Diabetes Care and Dexcom for in-kind donations to this investigator initiated study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 45 years of age (inclusive)
* A diagnosis of type 1 diabetes, as defined by Diabetes Canada, for at least 12 months
* A viable singleton pregnancy confirmed by ultrasound, less than 14 weeks gestation
* Currently on intensive insulin therapy (≥ 3 injections, or Continuous subcutaneous insulin infusion (CSII)
* Willingness to use the study devices throughout the trial
* A1c ≥ 6.2% and <10% measured any time during pregnancy prior to enrollment
* Able to provide informed consent
* Have access to email

Exclusion Criteria:

* Non-type 1 diabetes
* Current treatment with drugs known to interfere with glucose metabolism as judged by the investigator such as high dose systemic corticosteroids
* Known or suspected allergy to insulin
* Women with nephropathy (estimated glomerular filtration rate [eGFR] <45), severe autonomic neuropathy, uncontrolled gastroparesis or severe proliferative retinopathy, as judged by the investigator, that is likely to interfere with the normal conduct of the study and interpretation of study results
* Total daily insulin dose <8 or >250 units/day at screening
* Severe visual or hearing impairment, as judged by the investigator to impact treatment compliance
* Unable to communicate effectively in English or French as judged by the investigator
* Current use of Tandem Control IQ, DIY looping system, 670G in Auto Mode, or alternate closed-loop system as judged by the investigator
* Any reason judged by the investigator that would likely interfere with the normal conduct of the study and interpretation of study results

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Glycemic control as reflected by percent glucose time-in-range | 16 weeks until 34 weeks gestation
  Time in range (3.5 to 7.8 mmol/L) per day assessed by CGM glucose measurement

SECONDARY OUTCOMES:
Percent time spent above target range per day (+/-SD) | 16 weeks gestation until delivery of neonate
  Glucose above target range defined as glucose >7.8 mmol/L; Blood glucose will be assessed using CGM data
Percent time spent below target range per day (+/-SD) | 16 weeks gestation until delivery of neonate
  Glucose below target range defined as glucose < 3.5 mmol/L; Blood glucose will be assessed using CGM data
Mean blood glucose measurement at 24 and 34 weeks (+/-SD) | 24 and 34 weeks gestation
  Blood glucose measured in mmol/L and assessed using CGM data
Proportion of participants who experience maternal hypoglycemic events | 16 weeks gestation until delivery of neonate
  Maternal hypoglycemic events defined as ≥15 minutes with CGM glucose <3.5 mmol/L [level 1] or <2.8 mmol/L [level 2]; Blood glucose will be assessed using CGM data
Glycemic variability reflected by the coefficients of variation and standard deviations of CGM data | 16 weeks gestation until delivery of neonate
  Blood glucose measured in mmol/L and assessed using CGM data
Diabetes-related distress to the participant | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Diabetes-related distress will be assessed four times during the study using the Diabetes Distress Screening Scale (DDSS17)
Fear of hypoglycemia | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Fear of hypoglycemia will be assessed four times during the study using the Hypoglycemia Fear Survey Questionnaire II (HFSQ II)
Fear of hyperglycemia | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Fear of hyperglycemia will be assessed four times during the study using the g. Hyperglycemia Fear in Pregnancy Survey
Sleep quality | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Sleep quality will be assessed at four times during the study using the Modified Pittsburgh Sleep Quality Index (PSQI)
Health-related quality of life | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Health-related quality of life will be assessed four times during the study using the Euro Quality of life questionnaire (EQ-5D-5L)
Work productivity | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Work productivity will be assessed four times during the study using the Work Productivity and Activity Impairment survey
Diabetes-related distress to the partners | 7-13 weeks + 6 days gestation, 24 weeks gestation, 34 weeks gestation, 6 weeks postpartum
  Diabetes-related distress to the partners will be assessed four times during the study using the Partner Diabetes Distress Scale
Proportion of participants who experience preeclampsia events | 16 weeks gestation until delivery of neonate
  Preeclampsia is defined as pregnancy ≥20 wks gestation with SBP ≥140mmHg and/or DBP ≥90 mmHg on ≥2 occasions a minimum of 6 hrs apart and new-onset of proteinuria (defined as urinary excretion ≥0.3g protein on a 24-hr urine specimen, or ≥ 2+ by urinary dipstick, or ≥30mg protein/mmol of urinary creatinine by spot testing) OR ≥1 of the following adverse conditions:
  * Eclampsia (Seizures in pregnancy)
  * Elevated liver function tests (Increased AST and/or ALT >70 IU/L)
  * Decreased platelet count <100 x 109/L
  * Elevated serum creatinine (>80 μmol/L)
  * Small for gestational age infant (birth weight <10th percentile)
Proportion of participants who experience gestational hypertension events | 16 weeks gestation until delivery of neonate
  Gestational hypertension is defined as a woman ≥20 weeks gestation with a systolic blood pressure of ≥140 mm Hg and/or a diastolic blood pressure ≥90 mm Hg on ≥2 occasions a minimum of 6 hours apart without proteinuria
Proportion of participants who experience worsening chronic hypertension events | 16 weeks gestation until delivery of neonate
  Chronic hypertension is defined as hypertension that is present at <20 weeks gestation or pre-pregnancy
Proportion of participants who have caesarean deliveries | 16 weeks gestation until delivery of neonate
Proportion of participants who experience preterm births | Delivery of neonate to 6 weeks postpartum
  Preterm birth defined as birth occurring <37 weeks gestation
Proportion of babies born large for gestational age (>90th percentile) | Delivery of neonate
Proportion of babies born small for gestational age (<10th percentile) | Delivery of neonate
Mean neonatal birthweight (+/-SD) | Delivery of neonate
  Birthweight measured in kilograms
Comparison of birthweight z-score | Delivery of neonate
Proportion of babies born with neonatal hypoglycemia | Delivery of neonate
Proportion of neonates admitted to intensive care unit admission | Delivery of neonate to 6 weeks postpartum
  Admission to neonatal intensive care unit admission defined as admission of 24 hours or more
Proportion of participants who experienced pregnancy loss or miscarriage (< 20 weeks, stillbirth ≥20 weeks, neonatal loss up to 28 days) | 7-13 weeks until delivery of neonate + up to 28 days
Proportion of participants who experience episodes of severe hypoglycemia | 7-13 weeks + 6 days gestation until delivery of neonate
  Severe hypoglycemia defined as a hypoglycemic episode requiring assistance from another person.
Proportion of participants who experience episodes of diabetic ketoacidosis | 7-13 weeks + 6 days gestation until delivery of neonate
  Diabetic ketoacidosis (DKA) is defined as an episode with elevated plasma ketones which can be categorized as possible DKA (mild/ self- treated [plasma ketones 0.6 - 1.5mmol/L], moderate/self-treated (plasma ketones > 1.5mmol/L which resolves without hospital admission), or capillary blood ketones >3.0 mol/L without an anion gap of > 15 with admission to hospital for another reason [i.e. prevention of DKA]) or confirmed DKA (severe, with either plasma ketones > 3.0mmol/L or positive serum ketones with an anion gap (Na -(CI+HC03) > 15 and requiring hospital admission for IV fluids and IV insulin to correct the abnormal metabolic state).
Proportion of participants who experience device-related adverse events | 7-13 weeks + 6 days gestation until delivery of neonate
  Device-related adverse events include skin reactions and insulin delivery failures.

CONTACTS AND LOCATIONS:
Overall Officials: Lois Donovan, MD, Principal Investigator — University of Calgary; Denice Feig, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (14):
- Australia (5):
  - Campbelltown Hospital, Campbelltown
  - Royal Prince Alfred Hospital, Camperdown
  - Canberra Hospital, Garran
  - Royal Women's Hospital, Parkville
  - Westmead Hospital, Westmead
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - BC Women's Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Lawson Health Research Institute, London, Ontario
  - Sunnybrook, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University of Montreal - CHUM, Montreal, Quebec
  - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Persson M, Norman M, Hanson U. Obstetric and perinatal outcomes in type 1 diabetic pregnancies: A large, population-based study. Diabetes Care. 2009 Nov;32(11):2005-9. doi: 10.2337/dc09-0656. Epub 2009 Aug 12. PMID 19675195
- [Background] Feig DS, Hwee J, Shah BR, Booth GL, Bierman AS, Lipscombe LL. Trends in incidence of diabetes in pregnancy and serious perinatal outcomes: a large, population-based study in Ontario, Canada, 1996-2010. Diabetes Care. 2014 Jun;37(6):1590-6. doi: 10.2337/dc13-2717. Epub 2014 Apr 4. PMID 24705609
- [Background] Evers IM, de Valk HW, Visser GH. Risk of complications of pregnancy in women with type 1 diabetes: nationwide prospective study in the Netherlands. BMJ. 2004 Apr 17;328(7445):915. doi: 10.1136/bmj.38043.583160.EE. Epub 2004 Apr 5. PMID 15066886
- [Background] Murphy HR, Roland JM, Skinner TC, Simmons D, Gurnell E, Morrish NJ, Soo SC, Kelly S, Lim B, Randall J, Thompsett S, Temple RC. Effectiveness of a regional prepregnancy care program in women with type 1 and type 2 diabetes: benefits beyond glycemic control. Diabetes Care. 2010 Dec;33(12):2514-20. doi: 10.2337/dc10-1113. PMID 21115765
- [Background] Maresh MJ, Holmes VA, Patterson CC, Young IS, Pearson DW, Walker JD, McCance DR; Diabetes and Pre-eclampsia Intervention Trial Study Group. Glycemic targets in the second and third trimester of pregnancy for women with type 1 diabetes. Diabetes Care. 2015 Jan;38(1):34-42. doi: 10.2337/dc14-1755. Epub 2014 Nov 3. PMID 25368104
- [Background] Murphy HR, Bell R, Cartwright C, Curnow P, Maresh M, Morgan M, Sylvester C, Young B, Lewis-Barned N. Improved pregnancy outcomes in women with type 1 and type 2 diabetes but substantial clinic-to-clinic variations: a prospective nationwide study. Diabetologia. 2017 Sep;60(9):1668-1677. doi: 10.1007/s00125-017-4314-3. Epub 2017 Jun 8. PMID 28597075
- [Background] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Background] Tennant PW, Glinianaia SV, Bilous RW, Rankin J, Bell R. Pre-existing diabetes, maternal glycated haemoglobin, and the risks of fetal and infant death: a population-based study. Diabetologia. 2014 Feb;57(2):285-94. doi: 10.1007/s00125-013-3108-5. Epub 2013 Nov 29. PMID 24292565
- [Background] Singh H, Murphy HR, Hendrieckx C, Ritterband L, Speight J. The challenges and future considerations regarding pregnancy-related outcomes in women with pre-existing diabetes. Curr Diab Rep. 2013 Dec;13(6):869-76. doi: 10.1007/s11892-013-0417-5. PMID 24013963
- [Background] Singh H, Ingersoll K, Gonder-Frederick L, Ritterband L. "Diabetes Just Tends to Take Over Everything": Experiences of Support and Barriers to Diabetes Management for Pregnancy in Women With Type 1 Diabetes. Diabetes Spectr. 2019 May;32(2):118-124. doi: 10.2337/ds18-0035. PMID 31168282
- [Background] Langer N, Langer O. Pre-existing diabetics: relationship between glycemic control and emotional status in pregnancy. J Matern Fetal Med. 1998 Nov-Dec;7(6):257-63. doi: 10.1002/(SICI)1520-6661(199811/12)7:63.0.CO;2-H. PMID 9848689
- [Background] Berg M. Pregnancy and diabetes: how women handle the challenges. J Perinat Educ. 2005 Summer;14(3):23-32. doi: 10.1624/105812405X57552. PMID 17273439
- [Background] Berg M, Honkasalo ML. Pregnancy and diabetes--a hermeneutic phenomenological study of women's experiences. J Psychosom Obstet Gynaecol. 2000 Mar;21(1):39-48. doi: 10.3109/01674820009075607. PMID 10907214
- [Background] Gupton A, Heaman M, Cheung LW. Complicated and uncomplicated pregnancies: women's perception of risk. J Obstet Gynecol Neonatal Nurs. 2001 Mar-Apr;30(2):192-201. doi: 10.1111/j.1552-6909.2001.tb01535.x. PMID 11308109
- [Derived] Donovan LE, Lemieux P, Dunlop AD, Yamamoto JM, Murphy HR, Simmons D, Bell RC, Chaput KH, Benham JL, Ross GP, Nerenberg KA, Booth JE, Perkins BA, Mohammad K, Ntanda HN, King JA, Tomlinson G, Feig DS; CIRCUIT Collaborative Group. Closed-Loop Insulin Delivery in Type 1 Diabetes in Pregnancy: The CIRCUIT Randomized Clinical Trial. JAMA. 2025 Dec 23;334(24):2176-2185. doi: 10.1001/jama.2025.19578. PMID 41134589